CLINICAL TRIAL: NCT07084974
Title: Choosing a Trunk Assistance Exoskeleton: Issues of Cumulative Lumbar Loading, Muscle Fatigue, and Discomfort During Repetitive Lifting Tasks
Brief Title: Evaluation of Trunk Assistance Exoskeleton
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TOPMED (Other)
Collaborators: Institut de Recherche Robert-Sauvé en Santé et en Sécurité du Travail (Other); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 502_IRSST_Exo
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Exoskeleton Device
Keywords: exoskeleton; trunk assistance; cumulative lumbar load; muscular fatigue; lifting task; comfort; acceptability

STUDY DESIGN:
Intervention Model Description: All participants will begin by the adjustement and practice session. The order of the 4 other interventions(No trunk assistance, and the 3 exoskeletons: Uplift Lite, Biolift and Laevo Flex) will be randomized in between participants to reduce sequence effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Repeated measures intervention group (Experimental): Participants will perform 5 different intervention sessions:
  An adjustment and practice session which is always performed first, then participants will performed 4 lifting tasks sessions in randomized order:
  * No trunk assistance session
  * Uplift Lite exoskeleton session
  * Biolift exoskeleton session
  * Laevo Flex exoskeleton session
  During each lifting task session, participants will perform 3 blocks of 20 minutes of the lifting task. The lifting task is a box transfer tasks from the ground to a table adjusted at hip height. The task rythm is 7 cycles per minute. The box weight is equivalent to 10% of their maximal lifting strength. The handles of the box are positioned at 28 cm above the bottom of the box. Total session duration is about 3 hours for all sessions. Participants will have between 4 and 14 days of rest in between each sessions.
  Interventions: Device: Adjustment and practice session; Device: No trunk assistance; Device: Uplift Lite exoskeleton; Device: Biolift exoskeleton; Device: Laevo Flex exoskeleton

INTERVENTIONS:
Device: Adjustment and practice session — During the adjustment and practice session, participants will perform the lifting task with each exoskeleton after they are properly fitted. They will also perform the measurement sequence as to limit learning effects during lifting task sessions. The lifting task is a box transfer tasks from the ground to a table adjusted at the participant's hip height. The task rhythm is 7 cycles per minute. The box weight is equivalent to 10% of their maximal lifting strength. Total session duration is about 3 hours.
Device: No trunk assistance — This lifting task session is performed without any trunk assistance exoskeleton. Participants perform 3 blocks of 20 minutes of the lifting task. The lifting task is a box transfer tasks from the ground to a table adjusted at the participant's hip height. The task rhythm is 7 cycles per minute. The box weight is equivalent to 10% of their maximal lifting strength. Total session duration is about 3 hours.
Device: Uplift Lite exoskeleton — This lifting task session is performed with the Mawashi Uplift Lite trunk assistance exoskeleton. Participants will perform 3 blocks of 20 minutes of the lifting task. The lifting task is a box transfer tasks from the ground to a table adjusted at the participant's hip height. The task rhythm is 7 cycles per minute. The box weight is equivalent to 10% of their maximal lifting strength. Total session duration is about 3 hours.
Device: Biolift exoskeleton — This lifting task session is performed with the Biolift trunk assistance exoskeleton. Participants perform 3 blocks of 20 minutes of the lifting task. The lifting task is a box transfer tasks from the ground to a table adjusted at the participant's hip height. The task rhythm is 7 cycles per minute. The box weight is equivalent to 10% of their maximal lifting strength. Total session duration is about 3 hours.
Device: Laevo Flex exoskeleton — This lifting task session is performed with the Leavo Flex trunk assistance exoskeleton. Participants perform 3 blocks of 20 minutes of the lifting task. The lifting task is a box transfer tasks from the ground to a table adjusted at the participant's hip height. The task rhythm is 7 cycles per minute. The box weight is equivalent to 10% of their maximal lifting strength. Total session duration is about 3 hours.

SUMMARY:
The goal of this interventional study is to evaluate the effect of three different designs of trunk assistance exoskeletons on cumulative lumbar load, trunk extensors' muscular fatigue and comfort in healthy volunteers. The main questions it aims to answer is: will exoskeletons reduce muscle fatigue and cumulative lumbar load. Participants will :

* get each exoskeletons adjusted and then practice the lifting task and measurement sequence in a first session
* perform a lifting task for 4 blocks of 20 minutes on different sessions for each exoskeleton, another session is performed without assistance.

ELIGIBILITY:
Inclusion Criteria:

* Being able to communicate in french

Exclusion Criteria:

* Back pain in the last year
* Back pain for more than a week in the years prior
* Musculoskeletal injury in the last year
* Trunk musculoskeletal system surgery in the last year
* Scoliosis diagnostic
* Systemic illness, degenerative disease or syndrome related to the trunk musculoskeletal or nervous system
* Body mass index over 35 kg/m^2
* History of neurological damage
* Any contraindication to the practice of physical activity
* Incapacity to perform the lifting task at the specified rythm
* Medication with a negative impact on balance

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in spinal compression | For each lifting task session, change between session's baseline(immediately before the first lifting task block) and immediately after each lifting task block
  Stadiometer measurements require an electronic comparator (Mitutoyo; model 543-730B) mounted on a height-adjustable structure that allows alignment with the longitudinal axis of the spine. To measure spinal compression, the participant should position themselves face down against the wall, feet shoulder-width apart (template on the floor), knees fully extended, arms at their sides, and the following points in "light" contact with the wall: forehead, nose, pelvis (or navel), and toes (without shoes, with socks). The assessor will be asked to take the measurements (10 measurements) at the end of expiration, where they will be asked to hold their breath for 2-3 seconds. The baseline for the lifting task sessions is measured before all lifting task blocks. This measurement, expressed in millimeters, reflects only the vertical position of the electronic comparator. Measure = Mean after Block X - Session's baseline mean(before block 1).
Change in muscular exertion perception | For each lifting task session, change between session's baseline(immediately before the first lifting task block) and immediately after each lifting task block
  Participants score their muscular exertion perception in 5 muscle groups (quadriceps, hamstrings, hip extensors, lumbar extensors, thorax extensors) on the Borg CR-10 scale. The baseline for the lifting task sessions is measured before all lifting task blocks. There are 12 levels to this scale(Minimum=0(No exertion) maximum=10(maximal exertion), all integer values, 0.5 is also an option.
Change in maximal lifting strength | For each lifting task session, change between session's baseline(immediately before the first lifting task block) and immediately after the last lifting task block
  Maximal lifting strength is assessed by measuring pulling force on a bar at knee level with a strain gauge. The handle is held firmly by both hands. Participants were asked to bend at the hips and knees so as to keep an extended lower back during the trials, similar to a deadlifting position. During each trial, participants were asked to progressively pull harder on the bar without jerking for 5 seconds. The maximal value expressed in newtons during each trial was used. The baseline measurement is the mean of 3 trials with a 2 minute pause in between trials. Only 1 trial was performed after the last lifting block so as to better assess muscular fatigue by limiting time for recovery.

SECONDARY OUTCOMES:
Exoskeleton assistance score | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants scored the assistance they felt wearing an exoskeleton on a 5-level Likert scale(min: no assistance= 0, max: considerable assistance = 4).
Number of cycles with parasitic forces score | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants scored the estimated proportion of cycles where parasitic forces were experienced (min:0% of cycles=0 , max:100% of cycles=4) on a 5-level Likert scale.
Magnitude of parasitic forces score | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants scored the magnitude of parasitic forces when these were experienced (min: no forces experienced=0 , max: very high forces experienced=5) on a 6-level Likert scale.
Number of cycles with restriction of movement | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants scored the estimated proportion of cycles where the exoskeleton restrained their movement (min:0% of cycles=0 , max:100% of cycles=4) on a 5-level Likert scale.
Magnitude of restriction of movement | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants scored the magnitude of movement restrictions caused by the exoskeleton when these were experienced (min: no movement restriction experienced=0 , max: very high movement restrictions experienced=5) on a 6-level Likert scale.
Number of cycles with postural instability | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants scored the estimated proportion of cycles where the exoskeleton caused postural instability (min:0% of cycles=0 , max:100% of cycles=4) on a 5-level Likert scale.
Magnitude of postural instability | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants scored the magnitude of postural instability caused by the exoskeleton when these were experienced (min: no postural instability experienced=0 , max: very high postural instability experienced=5) on a 6-level Likert scale.
Exoskeleton pressure points score | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants scored the pressure points caused by the exoskeleton when these were experienced on a 5 item 7-level Likert scale(min: no pressure points experienced=0 , max: extreme pressure points experienced=6). The 5 items were different anatomical regions (thighs, hips/lower back, back of thorax, front of thorax, above the shoulders). Combined score is the sum of all items (min: no pressure points experienced=0 , max: extreme pressure points experienced=30).
Exoskeleton discomfort score | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants scored the discomforts caused by the exoskeleton when these were experienced on a 5 item 5-level Likert scale (min: strongly disagree=-2 , max: strongly agree=+2). The 5 items were different types of discomforts (being hot, sweatiness, itching or iritation of the skin, pinch point, pain). Combined score is the sum of all items (min: no discomforts experienced=-10 , max: extreme discomforts experienced=10).
Exoskeleton comfort score | For each lifting task session where the participant wore a trunk assistance exosqueleton, immediately after the last lifting task block
  Participants responded to the statement "I think this exoskeleton is comfortable" on a 5-level Likert scale (min: strongly disagree=-2 , max: strongly agree=+2).

CONTACTS AND LOCATIONS:
Locations (1):
- TOPMED, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No